CLINICAL TRIAL: NCT06944496
Title: A Phase III, Randomized Trial Comparing RC48 Plus Chemotherapy and Tislelizumab With Tislelizumab Plus Chemotherapy as First-line Treatment in Participants With HER2 Low Advanced Gastric or Gastrioesophageal Junction Adenocarcinoma (RC48-C039)
Brief Title: A Study of Disitamab Vedotin Combined With Tislelizumab and Chemotherapy Versus Tislelizumab Combined With Chemotherapy in HER2-Low Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RemeGen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C039
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Gastric Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tislelizumab combined with CAPOX (Active Comparator)
  Interventions: Biological: Tislelizumab+Oxaliplatin+Capecitabine
- Disitamab Vedotin Combined with Tislelizumab and CAPOX (Experimental)
  Interventions: Biological: Disitamab Vedotin+Tislelizumab+Oxaliplatin+Capecitabine

INTERVENTIONS:
Biological: Disitamab Vedotin+Tislelizumab+Oxaliplatin+Capecitabine — Disitamab Vedotin: 2.5 mg/kg, IV, D1, Q2W; Tislelizumab: 200 mg, IV, D1, Q3W Oxaliplatin: 100 mg/m², IV, D1, Q3W; Capecitabine: 750 mg/m², po, BID, D1-D14, Q3W
  Arms: Disitamab Vedotin Combined with Tislelizumab and CAPOX
Biological: Tislelizumab+Oxaliplatin+Capecitabine — Tislelizumab: 200 mg, IV, D1, Q3W Oxaliplatin: 130 mg/m², IV, D1, Q3W; Capecitabine: 1000 mg/m², po, BID, D1-D14, Q3W
  Arms: Tislelizumab combined with CAPOX

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of **Disitamab Vedotin combined with Tislelizumab and CAPOX versus Tislelizumab combined with CAPOX** as first-line treatment for patients with HER2-low advanced gastric or gastroesophageal junction adenocarcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily consent to participate in the study and sign the informed consent form
* Expected survival period >12 weeks
* ECOG Performance Status 0 or 1
* Histologically confirmed unresectable locally advanced, metastatic, or recurrent gastric or gastroesophageal junction adenocarcinoma
* No prior systemic therapy for locally advanced or metastatic gastric cancer
* HER2-low expression
* At least one assessable lesion according to RECIST v1.1 criteria
* Adequate organ function
* For female subjects: They should be surgically sterilized, postmenopausal, or agree to use a medically approved contraceptive method (such as an intrauterine device, contraceptive pill, or condom) during the study treatment period and for 6 months after the end of the study treatment. A blood pregnancy test must be negative within 7 days before the study medication is administered, and they must not be breastfeeding
* For male subjects: They should be surgically sterilized or agree to use a medically approved contraceptive method during the study treatment period and for 6 months after the end of the study treatment
* Able to understand the study requirements and willing to comply with the study and follow-up procedures

Exclusion Criteria:

* Presence of central nervous system (CNS) metastasis and/or carcinomatous meningitis
* Peripheral neuropathy > Grade 1
* Tumor lesions with a tendency to bleed
* Uncontrolled diarrhea
* Bone metastases with a risk of paraplegia
* Past or current interstitial lung disease, or presence of drug-induced pneumonia, radiation pneumonia, or severely impaired lung function
* Other malignancies within 5 years before the first dose, except for those expected to be cured with treatment (e.g., adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated with curative surgery)
* Pregnant or breastfeeding women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Estimated)
Dates: Start 2025-05-15 (Estimated); Primary Completion 2028-05-15 (Estimated); Study Completion 2030-05-15 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 24 months

SECONDARY OUTCOMES:
Overall Survival | up to 5 years
Objective Response Rate | 24 months
Disease Control Rate | 24 months
Duration of Response | 24 months
Patient-Reported Outcomes | 24 months
Adverse Events | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, BJ-Beijing, China